CLINICAL TRIAL: NCT01822925
Title: A Phase II Randomized, Double-Blind, Parallel Group, Dose-Ranging, Placebo-Controlled Study to Assess the Safety And Effectiveness Of DA-9801 in the Treatment of Subjects With Diabetic Neuropathy
Brief Title: Study of DA-9801 to Treat Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA9801-DN-001
Record Dates: First submitted 2013-03-21; First posted 2013-04-04 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetes; Pain; Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Pain | interventions — DA-9801

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DA-9801 300mg (Experimental): DA-9801 will be administered in tablet form, 100mg taken 3 times daily to subjects randomized to this arm of the study. Subjects will be expected to take this medication for 12 weeks.
  Interventions: Drug: DA-9801 300mg
- DA-9801 600mg (Experimental): DA-9801 will be administered in tablet form, 200 mg taken 3 times daily to subjects randomized to this arm of the study. Subjects will be expected to take this medication for 12 weeks.
  Interventions: Drug: DA-9801 600mg
- DA-9801 900mg (Experimental): DA-9801 will be administered in tablet form, 300 mg taken 3 times daily to subjects randomized to this arm of the study. Subjects will be expected to take this medication for 12 weeks.
  Interventions: Drug: DA-9801 900mg
- Placebo (Placebo Comparator): Placebo (same formulation as DA-9801 but without the active ingredients) will be administered in tablet form, 3 times daily to subjects randomized to this arm of the study. Subjects will be expected to take this tablet for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DA-9801 300mg — 300 mg of DA-9801 in tablet form, 100 mg to be taken 3 times daily for 12 weeks.
  Arms: DA-9801 300mg
Drug: DA-9801 600mg — 600 mg of DA-9801 in tablet form, 200 mg to be taken 3 times daily for 12 weeks.
  Arms: DA-9801 600mg
Drug: DA-9801 900mg — 900 mg of DA-9801 in tablet form, to be taken 300 mg to be taken 3 times daily for 12 weeks.
  Arms: DA-9801 900mg
Drug: Placebo — Placebo, in tablet form, to be taken 3 times daily for 12 weeks. The placebo is the same formulation as DA-9801 except that it does not contain the active pharmaceutical ingredient.
  Arms: Placebo

SUMMARY:
To evaluate the effectiveness of DA-9801 at 300mg, 600mg, 900mg and placebo, in reducing pain in subjects with diabetic neuropathic pain compared to their baseline values.

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel group, dose ranging, placebo-controlled study where eligible subjects (age 18 to 75 years) will have an average pain score ≥ 4 on an 11-point Likert numerical rating scale (NRS) for at least four days each week prior to randomization as assessed by daily pain diaries. Eligible subjects will be randomized to a 1:1:1:1 ratio to receive 300mg, 600mg, 900mg of DA-9801, or placebo three times a day for 12 weeks. During and at the end of the 12-week treatment period subjects will be evaluated for safety and efficacy parameters. A follow-up visit for safety will occur two weeks after the last treatment visit (TV).

The Screening Phase (2 weeks) is designed to determine whether subjects are eligible to proceed to the Treatment Phase of the study and consists of a series of screening assessments designed to determine eligibility. Eligible subjects will undergo a two-week washout period for medications and therapies administered for pain management.

At or up to 21 days before the Screening Visit, written informed consent from (ICF) the subject will be obtained by the Investigator or a suitably qualified designee before the performance of any protocol specific procedure. At the Screening Visit, the subject will be issued a daily diary in order to record daily pain level during the screening phase.

The Treatment Phase (TV0 to TV12) begins with a series of assessments designed to confirm the subjects' continued eligibility. The site will collect the daily diary and the subject's pain score will be determined. Only subjects whose average pain score is ≥ 4 for at least four days each week will be randomized to any of the four treatment groups.

DA-9801 administration schedule is three times per day, starting from TV0 to TV12.

During this study phase subjects will be evaluated on a weekly basis. Efficacy evaluations each week will include the subject's global impression of improvement and CGI of pain. Safety evaluations during the Treatment Phase will consist of adverse event assessments at each visit.

The Follow-up Visit (two weeks after last TV) The Follow-up Visit is designed to assess safety and will occur 14 days after the last TV. If the subject is withdrawn from the study prior to TV12, the subject should be exited from the study AFTER completing the specified assessments for that visit.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 to 75 years of age
* Diagnosed with Type I or Type II diabetes
* HbA1c ≤ 12% at the time of screening
* Has diabetic neuropathic pain (numbness, soreness, shooting or poking pain) in the lower extremities for more than 3 months prior to screening and with no adequate relief from other treatments
* Has an average pain score of ≥ 4 for 24 hours at least 4 days out of the week prior to randomization as assessed by the 11-point Likert NRS.
* If female of childbearing potential, subject must have a negative serum pregnancy test at screening
* Understands and is willing to participate in the clinical study and can comply with study procedures and visits.
* Normal cognitive and communicative ability as judged by clinical assessment and ability to complete self-reported questionnaires
* Subject is willing and able to give informed consent

Exclusion Criteria:

* Evidence of another type of neuropathic pain caused by a condition other than diabetes
* Pain from another source as severe or greater than the pain under study
* BMI (Body Mass Index) > 37 kg/m2
* Clinical signs of infection related to sores of any type on the legs
* Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding screening; or subject or physician anticipates use of any of these therapies by the subject during the course of the study
* Previous participation in the Treatment Phase of this Protocol
* History of drug or alcohol abuse, within the past 6 months
* Malignant disease not in remission for 5 years or more that has been medically or surgically treated without evidence of metastases
* Presence of one or more medical conditions, as determined by medical history, which seriously compromises the subject's ability to complete the study, including history of poor adherence with medical treatment, renal, hepatic, hematologic, active auto-immune or immune diseases that, in the opinion of the Investigator, would make the subject an inappropriate candidate for this study: c) One or more abnormal blood biochemistry analyte result that is ≥ 3 times that of the upper limit of the normal range; d) For laboratory results that are significantly lower than the normal range, specific criteria will be used to judge subject eligibility for randomization for Total protein, Albumin, and Hemoglobin or Platelets.
* Known history of having Acquired Immunodeficiency Syndrome (AIDS) or with a history known to be infected with Human Immunodeficiency Virus (HIV)
* New York Heart Association (NYHA) Class III and IV congestive heart failure (CHF), as defined by the following criteria: a)Class III: Symptoms with moderate exertion b)Class IV: Symptoms at rest
* Pregnant or breast feeding
* Women of child-bearing potential not using an effective birth control method. Women of child-bearing potential are defined as women physiologically capable of becoming pregnant, UNLESS they meet the following criteria:

  d) Post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels > 40mIU/m, OR; e) 6 weeks post surgical bilateral oophorectomy with or without hysterectomy, OR; f) Are using one or more of the following acceptable methods of contraception: surgical sterilization, hormonal contraception, and double-barrier methods. Reliable contraception should be maintained throughout the study and for 7 days after study discontinuation.
* Subjects with a diagnosis of psychiatric disorders such as major depressive disorder, bipolar disorder, obsessive compulsive disorder, generalized anxiety, dysthymia or suicidality/suicide ideation
* Administration of local anesthetic shot or systemic steroids within two months of screening
* Subjects not willing to undergo a two-week washout period for pharmacologic and non-pharmacologic pain management techniques

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Maislos, D.P.M, Principal Investigator — Houston Foot & Ankle Care
Locations (14):
- United States (14):
  - Center for United Research, Inc., Lakewood, California
  - Diablo Clinical Research, Walnut Creek, California
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - PAB Clinical Research, Brandon, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Novex Clinical Research, Inc., New Bedford, Massachusetts
  - Albany Medical Center, Albany, New York
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - KRK Research, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Houston Foot & Ankle Care, Houston, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Rainier Clinical Research Center, Inc., Renton, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 185 subjects were screened in this study from which, 128 subjects were randomized to the treatment groups, and 57 subjects were categorized as screen failure. Thirty-two (32) subjects were randomized to each of the four (4) study treatment groups: 900 mg DA-9801, 600 mg DA9801, 300 mg DA-9801 and placebo.
Groups:
- Placebo: Placebo oral tablets three (3) times per day.
- 300 mg DA-9801: 100 mg oral tablets three (3) times per day for total daily doses of 300 mg
- 600 mg DA-9801: 200 mg oral tablets three (3) times per day for total daily doses of 600 mg
- 900 mg DA-9801: 300 mg oral tablets three (3) times per day for total daily doses of 900 mg
Period: Overall Study
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Started | 32 | 32 | 32 | 32
Completed | 26 | 30 | 29 | 27
Not Completed | 6 | 2 | 3 | 5
Not completed — Adverse Event | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 2
Not completed — Taking prohibited medication | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 300 mg DA-9801: Oral tablets three (3) times per day for total daily doses of 300 mg
- 600 mg DA-9801: Oral tablets three (3) times per day for total daily doses of 600 mg
- 900 mg DA-9801: Oral tablets three (3) times per day for total daily doses of 900 mg
- Total: Total of all reporting groups
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801 | Total
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (8.8) | 59.7 (10.6) | 60 (10.6) | 61.6 (9.2) | 60.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 8 | 10 | 37
  Male | 22 | 23 | 24 | 22 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 6 | 7 | 21
  Not Hispanic or Latino | 29 | 27 | 26 | 25 | 107
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 6 | 7 | 4 | 22
  White | 24 | 25 | 24 | 28 | 101
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 32 | 32 | 128
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (3.9) | 30.8 (4.3) | 31.8 (3.5) | 31.2 (3.9) | 31 (3.9)
Height [Mean (Standard Deviation); unit: Inches] | 68.9 (4.6) | 69 (4.5) | 68.9 (4) | 69.4 (4.5) | 69 (4.4)
Weight [Mean (Standard Deviation); unit: lbs] | 205 (41.9) | 207 (35.4) | 217 (31.3) | 215 (41.2) | 211 (37.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinic Visit Pain Score at the 12 Week Visit Compared to Baseline as Assessed by the 11-point Likert Numerical Rating Scale (NRS)
Description: Pain score was assessed by the subject using the 11-point Likert rating scale for pain (0=no pain to 10=worst possible pain) prior to conduct of any other study assessment. The change in clinic visit pain score at the 12-week visit was compared to baseline.
Time Frame: Baseline to 12 weeks of treatment
Population: Intent-to-Treat (ITT) population - defined as all subjects who were randomized and had an ICF. The ITT population was the primary population for the analysis of primary and secondary endpoints.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
Scores on a scale
  TV 0 (Baseline) | 6.2 (1.93) | 6.6 (1.43) | 6.6 (1.54) | 6.5 (1.54)
  TV 12 | 4 (2.58) | 3.4 (2.49) | 3.5 (2.63) | 3.8 (2.69)

2. Secondary Outcome: Percentage Change in Clinic Visit Pain Score at the 12-week Visit Compared to Baseline as Assessed by the 11-point Likert Numerical Rating Scale (NRS)
Description: Pain intensity was assessed by the subject before any other protocol procedures at baseline and at the 12- week visit using an 11-point Likert-type numerical rating scale for pain (0=no pain, to 10=worst possible pain) (Negative values indicate percentage reductions).
Time Frame: Baseline and over 12 week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
Percentage change | -35.6 (35.3) | -45 (42) | -47 (36.5) | -41.4 (41.2)

3. Secondary Outcome: Number of Participants With at Least 30% Improvement Compared to Baseline as Assessed by the 11- Point Likert Numerical Rating Scale (NRS) at the Week 12 Clinic Visit
Description: Pain intensity was assessed by the subject before any other protocol procedures at baseline and week 12 based on 11-point Likert-type numerical rating scale for pain (0=no pain, to 10=worst possible pain).
  The number of participants who had achieved ≥ a 30% reduction in pain from the baseline was to be compared between the treatment groups and placebo.
Time Frame: Baseline to 12 week treatment period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 16 | 20 | 21 | 17

4. Secondary Outcome: Difference in Average Weekly Pain Score Between Dose Groups as Assessed by Daily Diary
Description: Average 24-hour pain intensity was assessed daily based on the 11-point Likert-type numerical rating scale for pain (0=no pain, to 10=worst possible pain). Average weekly pain scores are defined as 7* [(Pain Day 1 + Pain Day 2 + …+ Pain Day n)]/n where n is the number of available diary entries for the week. The minimum pain score for a week would be 0 and the maximum would be 70.
  Difference in the average weekly pain score at Week 12 is the score for each week minus the baseline .
Time Frame: Baseline to 12 week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Average weekly group pain score
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
Average weekly group pain score | 14.3 (13) | 19.8 (16.3) | 17.9 (18.1) | 15.9 (14.4)

5. Secondary Outcome: Difference in Average Weekly Most Severe Pain Score Between Dose Groups as Assessed by Daily Diary
Description: Most severe 24-hour pain intensity was assessed daily based on the 11-point Likert-type numerical rating scale for pain (0=no pain, to 10=worst possible pain). Average weekly most severe pain scores are defined as 7* [(Pain Day 1 + Pain Day 2 + …+ Pain Day n)]/n where n is the number of available diary entries for the week. The minimum possible pain score for a week would be 0 and the maximum possible would be 70.
  Difference in the average weekly pain score at Week 12 is the score at each week minus baseline .
Time Frame: Baseline to 12 week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weekly most severe pain score
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
weekly most severe pain score | 16 (14.7) | 23.2 (17.3) | 19.7 (19.6) | 18.9 (15.9)

6. Secondary Outcome: Difference in Average Weekly Overnight Pain Score Between Dose Groups as Assessed by Daily Diary
Description: Overnight pain intensity was assessed daily based on the 11-point Likert-type numerical rating scale for pain (0=no pain, to 10=worst possible pain). Average weekly overnight pain scores are defined as 7* [(Pain Day 1 + Pain Day 2 + …+ Pain Day n)]/n where n is the number of available diary entries for the week. The minimum possible pain score for a week would be 0 and the maximum possible would be 70.
  Difference in the average weekly overnight pain score at Week 12 is the score at each week minus baseline
Time Frame: Baseline to 12 week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average weekly overnight pain score
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
average weekly overnight pain score | 14.3 (14) | 19.9 (16.4) | 19 (18.1) | 16.9 (15.5)

7. Secondary Outcome: Change From Baseline Within Group- Difference in Average Weekly Pain Score Compared to Baseline as Assessed by Daily Diary
Description: Average weekly pain intensity was assessed daily based on the 11-point Likert-type numerical rating scale for pain (0=no pain, to 10=worst possible pain). Average weekly pain scores are defined as 7* [(Pain Day 1 + Pain Day 2 + …+ Pain Day n)]/n where n is the number of available diary entries for the week. The minimum possible pain score for a week would be 0 and the maximum possible would be 70.
  Difference in the average weekly pain score at Week 12 is the score at each week minus baseline.
Time Frame: Baseline to 12 week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average weekly pain score
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
average weekly pain score
  Baseline | 42.7 (10.7) | 45.9 (9.1) | 46.3 (10) | 44.2 (11.3)
  Week 12 | 28.3 (16.8) | 26.1 (17.1) | 28.4 (18.1) | 28.3 (18.5)
  Change | 14.3 (13) | 19.8 (16.3) | 17.9 (18.1) | 15.9 (14.4)

8. Secondary Outcome: Change From Baseline Within Group-Difference in Average Weekly Overnight Pain Score Compared to Baseline as Assessed by Daily Diary
Description: as for outcome 6
Time Frame: Baseline to 12 week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average weekly overnight pain score
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
average weekly overnight pain score
  Baseline | 43.7 (11) | 44.4 (11.8) | 46.5 (9.38) | 46.4 (12.6)
  Week 12 | 29.4 (17) | 24.5 (15.6) | 27.5 (19) | 29.5 (19.4)
  Change | 14.3 (14) | 19.9 (16.4) | 19 (18.1) | 16.9 (15.5)

9. Secondary Outcome: Number of Participants Considered to be Responders on Global Impression of Improvement (PGI-I) at Week 12
Description: PGI measures the subject's overall improvement in pain. The assessment was to be completed each week during the Treatment Phase.
  Global impression of improvement was assessed by the subject based on a 7 point scale (1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, 7-very much worse.
  Responders are defined as subjects with response of "very much improved", "much improved" or "minimally improved"
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 18 | 20 | 22 | 16

10. Secondary Outcome: Number of Participants Number of Participants Considered to be Responders in Clinical Global Impression (CGI) at Week 12
Description: CGI measures global severity of illness at a given point of time and the improvement from baseline. The assessment was to be completed by the Investigator at baseline and each week during the treatment phase.
  CGI responders were defined as subjects achieving a score of: (1): Very much improved or (2): Much improved or (3): Minimally improved on the clinician-rated CGI global improvement item.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 19 | 24 | 24 | 21

11. Secondary Outcome: Average Weekly Rescue Medication Use
Description: During the Treatment Periods, subjects taking 500 mg acetaminophen or Tylenol® for severe pain recorded the frequency and dosage in the daily diary. The use of 500 mg acetaminophen or Tylenol® was recorded for Morning, Afternoon or Evening time. For each subject, the total weekly rescue medication was calculated, and it was used to assess average weekly rescue medication use.
Time Frame: Week 1 to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Number analyzed (Participants) | 32 | 32 | 32 | 32
mg
  Week 1 | 1688 (3941) | 1469 (3617) | 1625 (4849) | 2141 (5008)
  Week 2 | 1844 (4683) | 1547 (3927) | 2156 (5566) | 2375 (5414)
  Week 3 | 1438 (3656) | 1391 (4666) | 1188 (3963) | 1063 (2602)
  Week 4 | 1313 (4484) | 563 (1384) | 531 (1905) | 625 (1535)
  Week 5 | 1047 (3817) | 844 (2807) | 375 (1621) | 578 (2703)
  Week 6 | 1078 (3612) | 859 (3114) | 172 (577) | 578 (2254)
  Week 7 | 1156 (3775) | 906 (3254) | 78.1 (314) | 891 (2999)
  Week 8 | 1156 (3971) | 719 (3976) | 93.8 (390) | 578 (1627)
  Week 9 | 1297 (4275) | 625 (2362) | 125 (707) | 500 (1827)
  Week 10 | 1438 (4499) | 1281 (4447) | 93.8 (530) | 531 (2359)
  Week 11 | 1266 (4076) | 891 (3184) | 109 (619) | 516 (2256)
  Week 12 | 1641 (5448) | 1109 (3638) | 93.8 (390) | 344 (1125)

ADVERSE EVENTS:
Time Frame: Treatment-Emergent Adverse Events (TEAEs) started on or after the first randomized study treatment administration and monitored for 14 weeks through study completion.
Arm/Group | Placebo | 300 mg DA-9801 | 600 mg DA-9801 | 900 mg DA-9801
Serious Adverse Events (participants affected / at risk) | 3/32 | 0/32 | 2/32 | 0/32
Other Adverse Events (participants affected / at risk) | 14/32 | 21/32 | 16/32 | 8/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | 300 mg DA-9801 (N=32) | 600 mg DA-9801 (N=32) | 900 mg DA-9801 (N=32)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | 300 mg DA-9801 (N=32) | 600 mg DA-9801 (N=32) | 900 mg DA-9801 (N=32)
Constipation (Gastrointestinal disorders) | 0 | 1 | 4 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Oedema peripheral (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 4 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Headache (Nervous system disorders) | 2 | 2 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No